CLINICAL TRIAL: NCT06702137
Title: The Effects of EXOPULSE Mollii Suit on Motor Functions in Patients With Multiple Sclerosis (EXOSEP Study)
Brief Title: EXOPULSE Mollii Suit, Motor Function & Multiple Sclerosis
Acronym: EXOSEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut De La Colonne Vertebrale Et Des Neurosciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-A00231-42
Record Dates: First submitted 2024-11-02; First posted 2024-11-22 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis
Keywords: Spasticity; Motor Functions; Quality of life
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: It is a randomized, controlled, double-blind, and cross-over study. Phase 1 is a randomized, controlled, double-blind, and cross-over study. In this phase, each participant will be randomly assigned to receive one session of active stimulation and one session of sham stimulation using the EXOPULSE Mollii suit (phase 1).
  The crossover design is appropriate for assessing symptomatic treatment of this chronic and relatively stable disease. Furthermore, the sessions will be separated by a wash-out interval of two weeks. Thus, a 2-week washout period should be enough to prevent a potential carry-over effect.
  At the end of phase 1 (two weeks after the second session of active or sham), an open-label phase (phase 2) will be proposed for all patients and will consist of 4 weeks of active stimulation (every other day stimulations for a total of 14 sessions).
  In total, each participant will be included in the study for 8 weeks (4 weeks for phase 1 and 4 weeks for phase 2).
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Condition (Active Comparator): Active sessions will last 1 hour each. The following parameters will be used for electric stimulation: low frequency (20 Hz), low current intensity (2 mA), with a small pulse width of 25-170 microseconds. These parameters were previously found to be safe in human studies. Based on the clinical exam of each patient, the spastic muscles will be targeted. EXOPULSE Mollii Suit is used for the activation of weak muscles or relaxation of spastic muscles mediated by a physiological reflex mechanism referred to as reciprocal inhibition. By sending an electrical signal to an antagonistic muscle, the spastic muscle will subsequently relax.
  Interventions: Device: EXOPULSE MOLLII SUIT (active)
- Control Condition (Sham Comparator): In the control condition, the patients will receive a sham stimulation, for which the control unit will be programmed to start stimulating for 1 minute then it will shut off. There is no risk related to the sham intervention since it consists of applying the same parameters used for the active session (low frequency: 20 Hz; current intensity: 2 mA; pulse width ranging from 25 to 170 µs) but for a shorter duration of time (1 minute instead of 1 hour).
  Interventions: Device: EXOPULSE MOLLII SUIT (sham)

INTERVENTIONS:
Device: EXOPULSE MOLLII SUIT (active) — This study aims to evaluate the effects of the EXOPULSE Mollii suit, a non-invasive assistive device that delivers transcutaneous electrostimulation. The suit includes a CE-labeled class IIa control unit and class I body garments. Equipped with 58 electrodes, the full-body suit stimulates various muscle groups to reduce spasticity by activating antagonistic muscles through reciprocal inhibition, rather than causing muscle contractions. Designed to relax spastic muscles, improve range of motion, prevent atrophy, enhance circulation, and provide pain relief, the device is easy to use, requiring only one hour of daily wear, with effects lasting over 24 hours.
  Current treatments for spasticity, such as botulinum toxin and oral medications, have limitations like side effects and minimal mobility improvement. The EXOPULSE Mollii suit offers an innovative alternative, with early studies indicating positive impacts on mobility and motor function.
  Arms: Experimental Condition
Device: EXOPULSE MOLLII SUIT (sham) — In the sham condition, the control unit will be programmed to start stimulating for 1 minute then it will shut off.
  Arms: Control Condition

SUMMARY:
Spasticity is a frequent and debilitating symptom in patients with multiple sclerosis (MS). It can alter the patients' balance, mobility, as well as their quality of life. The available therapeutic strategies for treating spasticity and related symptoms are usually faced with limited efficacy and numerous side effects.

For these reasons, non invasive stimulation techniques, namely transcutaneous stimulation by means of EXOPULSE Mollii suit, might be of help in this context.

DETAILED DESCRIPTION:
The investigators designed a randomized crossover, sham-controlled, double blind trial to demonstrate the improvement of motor functions and MS related symptoms following a single session of "active" versus "sham" EXOPULSE Mollii suit. A 2-week washout period should be enough to prevent a potential carry over effect. Two weeks after the end of this phase (phase 1), a second phase of this trial, an open label phase, will be proposed for all patients to understand the effects of EXOPULSE Mollii suit employed over four weeks (a session every other day for a total of 14 sessions) on MS related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Definite MS diagnosis according to the 2017 McDonald criteria since at least one month.
* Age between 18 and 75 years.
* Ability to walk freely or with the need of support (expanded disability status scale score (EDSS) < 7).
* Being free of relapses in the last three months.
* Being French speaker, able to understand verbal instructions, and affiliated to the national health insurance (sécurité sociale).
* Having spasticity with a score of at least 1+ on the MAS.
* Having a BBS score ≤46 associated in the literature with a risk of fall

Exclusion Criteria:

* Being included in another research protocol during the study period.
* Inability to undergo medical monitoring for the study purposes due to geographical or social reasons.
* Having a cardiac stimulator, a ventriculoperitoneal shunt, an intrathecal baclofen pump or other contraindications to using EXOPULSE Mollii suit.
* Being pregnant.
* Having a change in their pharmacological therapy in the last three months.
* Suffering from other somatic or neuropsychiatric diagnoses (e.g., arrhythmias, uncontrolled epilepsy, diseases causing osteoarticular and muscular pain).
* Having a body mass index above 35 Kg/m2.
* In case of the introduction of a medical device other than EXOPULSE Mollii suit during the study period
* Patients under juridical protection (" mesure de protection judiciare : tutelle, curatelle, sauvegarde de justice ")
* Prisoners.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
Improvement in balance using the BBS (Berg Balance Scale) ) | BBS will be evaluated at Day 1 (before & after the intervention, phase 1) and at Day 15 (before & after the intervention, phase 1)
  Balance will be assessed using the 14-item Berg Balance Scale (BBS) which has good psychometric properties in PwMS (concurrent validity, interrater reliability). The scale rates the balance using 56 points, with higher scores indicating better balance abilities. A score equal to or below 45 is commonly associated with the risk of falls across the literature.

SECONDARY OUTCOMES:
Assessment of the cumulative effects of EXOPULSE Mollii suit on balance using the BBS (Berg Balance Scale) after 4 weeks of using Exopulse Molii Suit | BBS evaluation will occur at Day 30 (before phase 2) and at Day 60 (at the end of phase 2)
  BBS has good psychometric properties in PwMS (concurrent validity, interrater reliability). The scale rates the balance using 56 points, with higher scores indicating better balance abilities. A score equal to or below 45 is commonly associated with fall risk across the literature.
Assessment of the spasticity using the MAS (Modified Ashworth Scale) | Spasticity according to MAS will be assessed through study completion at Day 1 (before and after the intervention, phase 1), at Day 15 (before and after the intervention, phase 1), at Day 30 (before phase 2) and at Day 60 (at the end of phase 2)
  Spasticity will be evaluated by examiners using the MAS (Modified Ashworth Scale)
Assessment of the spasticity using the VAS spasticity (Visual Analogue Scale) | VAS spasicity will be assessed through study completion at Day 1 (before and after the intervention, phase 1), at Day 15 (before and after the intervention, phase 1), at Day 30 (before phase 2) and at Day 60 (at the end of phase 2)
  Spasticity will be evaluated by patients using a VAS (Visual Analogue Scale)
Mobility will be assessed using the TUG (Time Up and Go) | Mobility according to TUG will be assessed through study completion at Day 1 (before and after the intervention, phase 1), at Day 15 (before and after the intervention, phase 1), at Day 30 (before phase 2) and at Day 60 (at the end of phase 2)
  The TUG is a validated test that assesses walking in PwMS (Bennett et al., 2017). The score is expressed as the time (in seconds) required to perform sequential motor tasks (standing up from the chair, walking to the line on the floor at a normal pace, turning, walking back to the chair at a normal pace, and finally sitting down).
Mobility will be assessed using the FES-I (Falls Efficacy Scale-International scale) | FES-I will be assessed at Day 30 (before phase 2) and at Day 60 (at the end of phase 2)
  Subjective risk of fall will be assessed using the French version of the Falls Efficacy Scale-International scale (FES-I) ; a 14-item scale that assesses the perceived risk of falling.
Mobility will be assessed using the MSWS-12 (Multiple Sclerosis Walking Scale - 12) | MSWS-12 will be assessed at Day 30 (before phase 2) and at Day 60 (at the end of phase 2)
  Subjective changes in walking would be evaluated by the Multiple Sclerosis Walking Scale - 12 (MSWS-12), a 12-item scale that examines the impact of MS on walking capacity, is a validated patient-reported measure for exploring this outcome.
Quality of life will be measured using the MusiQoL (Multiple Sclerosis International Quality of Life Questionnaire) | MusiQOL will be assessed at Day 30 (before phase 2) and at Day 60 (at the end of phase 2)
  This variable will be measured using the 31-item Multiple Sclerosis International Quality of Life Questionnaire (MusiQoL), which has good psychometric properties and yields a total score and subscores for nine dimensions: activity of daily living, psychological well-being, symptoms, friends' relationships, family relationships, satisfaction with health care, sentimental and sexual life, coping and rejection.
Pain will be assessed using a VAS (Visual Analogue Scale) | Pain according to VAS will be assessed through study completion at Day 1 (before and after the intervention, phase 1), at Day 15 (before and after the intervention, phase 1), at Day 30 (before phase 2) and at Day 60 (at the end of phase 2)
  VAS is a 10 mm straight horizontal line with one end meaning no pain and the other end meaning the worst pain imaginable
Fatigue will be assessed using a VAS (Visual Analogue Scale) | Fatigue according to VAS be assessed through study completion at Day 1 (before and after the intervention, phase 1), at Day 15 (before and after the intervention, phase 1), at Day 30 (before phase 2) and at Day 60 (at the end of phase 2)
  VAS is a 10 mm straight horizontal line with one end meaning no fatigue and the other end meaning extreme fatigue
Evaluation of overall improvement using the CGI (Clinical Global Impression) | CGI will be assessed at Day 1 (after the intervention, phase 1), at Day 15 (after the intervention, phase 1) and at Day 60 (at the end of phase 2)
  It consists of 7-point scale ranging from "very much improved since the initiation of treatment" to "very much worse since the initiation of treatment" (from 1 to 7)
Evaluation of patient's blinding to the type of stimulation in the crossover trial | Blinding wil be assessed at Day 1 (after the intervention) and at Day 15 (after the intervention) during Phase 1.
  This blind evaluation will be done in phase 1 using a dedicated questionnaire (only for each treatment condition, since all patients will receive the same active treatment in open phase 2).

CONTACTS AND LOCATIONS:
Overall Officials: Samar S AYACHE, MD, PhD, Principal Investigator — Clinical Neurophysiology department, Henri Mondor Hospital, Creteil, France
Locations (1):
- Clinical Neurophysiology Department, Henri Mondor Hospital, Créteil, VAL DE MARNE, France

REFERENCES:
- [Derived] Ayache SS, Mattar JG, Creange A, Abdellaoui M, Zedet M, Lefaucheur JP, Megherbi H, Khaled H, Abi Lahoud GN, Chalah MA. The effect of the EXOPULSE Mollii suit on motor functions in patients with multiple sclerosis - a randomized sham-controlled crossover trial. Mult Scler J Exp Transl Clin. 2025 Jun 19;11(2):20552173251348304. doi: 10.1177/20552173251348304. eCollection 2025 Apr-Jun. PMID 40547078